CLINICAL TRIAL: NCT02857348
Title: A Randomized Controlled Trial of a Video Game Intervention to Recalibrate Physician Heuristics
Brief Title: A Trial of a Video Game Intervention to Recalibrate Physician Heuristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Deepika Mohan, MD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO16070572
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Wounds and Injuries
Keywords: decision making; heuristics
MeSH Terms: conditions — Wounds and Injuries | interventions — Shift Work Schedule

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adventure video game (Experimental): Physicians in this arm of the trial will be asked to play Night Shift, an adventure video game, for one hour.
  Interventions: Behavioral: Night Shift
- Educational Module (Active Comparator): Physicians in this arm of the trial will be asked to use myATLS, an app designed by the American College of Surgeons to serve as an adjunct to the ATLS course, and Trauma Life Support MCQ Review, an app designed to help students prepare for the ATLS exam. They will be asked to spend at least one hour on the combined tasks.
  Interventions: Behavioral: Educational Module

INTERVENTIONS:
Behavioral: Night Shift — Night Shift is an adventure video game with the transformational goal of teaching physicians key characteristics of patients with non-representative severe injuries - injuries classified by the American College of Surgeons as life-threatening or critical but that do not fit the archetype of injuries typically requiring treatment at a trauma center. Players take on the persona of Andy Jordan, a young emergency physician who moves home after the disappearance of his estranged grandfather (Robert Jordan) and takes up a job in the local Emergency Department (ED). In the preamble, players learn they have two explicit objectives. First, they must diagnose and treat patients who present to their ED. Second they must solve the mystery of Robert's disappearance: was he murdered or has he simply chosen to disappear?
  Arms: Adventure video game
Behavioral: Educational Module — The educational module consists of two separate apps, both commercially available. myATLS includes a review of each chapter of the Advanced Trauma Life Support (ATLS) textbook, a series of videos demonstrating common trauma procedures, and clinical resources including checklists for use at the bedside. Trauma Life Support MCQ Review includes 550 multiple-choice questions with correct answers and explanations. The investigators will ask physicians to review the myATLS app and then complete questions in the Trauma Life Support MCQ Review, spending at least 1 hour on the combined tasks.
  Arms: Educational Module

SUMMARY:
The objective of this study is to compare the efficacy of a video game designed to recalibrate physician heuristics in trauma triage with a standard educational program.

DETAILED DESCRIPTION:
Treatment at trauma centers improves outcomes for patients with moderate-to-severe injuries. Accordingly, professional organizations, state authorities, and the federal government have endorsed the systematic triage and transfer of these patients to trauma centers either directly from the field or after evaluation at a non-trauma center. Nonetheless, between 30 to 40% of patients with moderate-to-severe injuries still only receive treatment at non-trauma centers, so-called under-triage. Most of this under-triage occurs because of physician decisions (rather than first-responder decisions). Existing efforts to change physician decision making focus primarily on knowledge of clinical practice guidelines and attitudes towards the guidelines. These strategies ignores the growing consensus that decision making reflects both knowledge as well as intuitive judgments (heuristics). Heuristics, mental short cuts based on pattern recognition, drive the majority of decision making. The investigators have developed an adventure video game (Night Shift) to serve as a novel method of recalibrating physician heuristics in trauma triage and will compare its efficacy with a standard educational program.

ELIGIBILITY:
Inclusion Criteria:

* Physicians who care for adult patients in the Emergency Department.
* Physicians who work at a non-trauma center.
* Physicians who work at a Level III/IV trauma center.

Exclusion Criteria:

* Physicians who work at a Level I/II trauma center.
* Physicians who do not practice in the US.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Under-triage rate | After completion of the intervention
  Physicians in both arms of the study will be randomized to complete one of two versions of a virtual simulation: a control version and a cognitive load version. They will complete the simulation upon completion of the intervention, ideally within one month of enrollment.
  The virtual simulation replicates the environment of the ED. Physicians have to manage 10 patients that appear concurrently, while also responding to a series of audio-visual distractors. Specifically, they must provide information on whether they will admit, transfer, or discharge the patients home. The investigators will calculate an under-triage rate for each physician (the number of simulated patients with severe injuries not transferred to a trauma center), summarize the under-triage rate by group (Night Shift v. educational control), and will compare the difference in those rates.

SECONDARY OUTCOMES:
The effect of cognitive load on the under-triage rate | After completion of the intervention
  As described above, participants will complete either a control or cognitive load version of the virtual simulation upon completion of the intervention, ideally within one month of the enrollment. As a secondary outcome measure, the investigators will assess the difference in under-triage rates of physicians who complete the simulation under control and cognitive load conditions, by intervention type.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Mohan, MD, Principal Investigator — University of Pittsburgh

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available on application to the investigator team.

REFERENCES:
- [Derived] Mohan D, Rosengart MR, Fischhoff B, Angus DC, Wallace DJ, Farris C, Yealy DM, Barnato AE. Using incentives to recruit physicians into behavioral trials: lessons learned from four studies. BMC Res Notes. 2017 Dec 28;10(1):776. doi: 10.1186/s13104-017-3101-z. PMID 29282154
- [Derived] Mohan D, Farris C, Fischhoff B, Rosengart MR, Angus DC, Yealy DM, Wallace DJ, Barnato AE. Efficacy of educational video game versus traditional educational apps at improving physician decision making in trauma triage: randomized controlled trial. BMJ. 2017 Dec 12;359:j5416. doi: 10.1136/bmj.j5416. PMID 29233854
- [Derived] Mohan D, Rosengart MR, Fischhoff B, Angus DC, Farris C, Yealy DM, Wallace DJ, Barnato AE. Testing a videogame intervention to recalibrate physician heuristics in trauma triage: study protocol for a randomized controlled trial. BMC Emerg Med. 2016 Nov 11;16(1):44. doi: 10.1186/s12873-016-0108-z. PMID 27835981